CLINICAL TRIAL: NCT02450812
Title: URANIS -Data Collection in Urological Centers During Treatment With Ra-223 Dichloride (Xofigo) Within the Framework of a Non-interventional Study Assessing Overall Survival (OS) and Effectiveness Predictors of Ra-223 Dichloride Treated mCRPC Patients in a Real Life Setting in Germany.
Brief Title: Non-interventional Study With Ra-223 Dichloride Assessing Overall Survival and Effectiveness Predictors for mCRPC Patients in a Real Life Setting in Germany
Acronym: URANIS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18043; XF 1503 (Other: NIS); EUPAS24796 (Other: ENCePP)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: mCRPC
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radium-223-dichloride (Xofigo, BAY88-8223): patients with mCRPC with symptomatic bone metastases
  Interventions: Drug: Radium-223-dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223-dichloride (Xofigo, BAY88-8223) — according to Summary of Product Characteristics

SUMMARY:
This observational prospective single arm cohort study is designed to assess overall survival, symptomatic skeletal event free survival and quality of life of metastatic Castration Resistant Prostate Cancer (mCRPC) patients receiving Radium- 223 under real life conditions. In addition, time to next tumor treatment (TTNT), mobility, quality of life and selfcare, independence in activities of daily living and safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male patients diagnosed with castration resistant adenocarcinoma of the prostate (CRPC) with symptomatic bone metastases without known visceral metastases
* Decision to initiate treatment with Radium-223 was made as per investigator's routine treatment practice

Exclusion Criteria:

-Patients participating in an investigational program with interventions outside of routine clinical practice and also in all non-interventional studies focusing on Radium- 223-dichloride.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of mCRPC patients with symptomatic bone metastases without known visceral metastases for whom the attending physician decided according to his/her medical practice to treat the patient with Radium-223 dichloride.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 60 months

SECONDARY OUTCOMES:
Evaluation of symptomatic skeletal event free survival (SSE-FS) of mCRPC patients | Up to 60 months
Estimation of the incidence of pathological fractures. | Up to 60 months
Time to next tumor treatment(s) (TTNT) | Up to 24 months
Incidence of treatment-emergent adverse events (TEAE) | Up to 30 days after last administration of Radium-223
Quality of life as patient reported outcome estimated using Functional Assessment of Cancer Therapy - Prostate (FACT-P) questionnaire | Up to 60 months
  The FACT-P questionnaire version 4 is a 39-item questionnaire consisting of five domains; 'Physical well-being', 'Social/Family well-being', 'Emotional well-being', 'Functional well-being' and 'Additional concerns' (consisting of items relating specifically to prostate cancer and/or its treatment) and uses a 0-4 Likert-scale.
Activities of daily living assessed according to the Katz-Index | Up to 7 months
Body function assessed in dimensions of "mobility", "self-care" and "domestic life" using the Medical Oncology Status in Europe Survey (MOSES) questionnaire | Up to 7 months
Estimation of the non-pathological fractures | Up to 60 months
Estimation of the bone associated events | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/